CLINICAL TRIAL: NCT04335968
Title: Melatonin for Prevention of Postoperative Delirium After Lower Limb Fracture Surgery in Elderly Patients: a Randomized Controlled Trial
Brief Title: Melatonin for Prevention of Postoperative Delirium After Lower Limb Fracture Surgery in Elderly Patients
Acronym: DELIRLESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APHP180594
Record Dates: First submitted 2020-02-28; First posted 2020-04-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Orthopedic Surgery
Keywords: delirium; aging; Perioperative neurocognitive disorders; melatonine; orthopedic surgery
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Prospective, national multicentric (21 centers), phase III, superiority, comparative randomized (1:1) double-blinded clinical trial with two parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): melatonin 4mg per os every night, starting the evening before surgery (or 2 hours before emergency surgery) and until day 5 after surgery
  Interventions: Drug: Melatonin 4 mg
- Control group (Placebo Comparator): placebo of this drug with the same schedule, during the same period of time.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Melatonin 4 mg — melatonin 4mg per os every night, starting the evening before surgery (or 2 hours before emergency surgery) and until day 5 after surgery.
  Arms: Experimental group
Drug: Placebo oral tablet — placebo of this drug with the same schedule, during the same period of time.
  Arms: Control group

SUMMARY:
Postoperative delirium (POD) is one of the most frequent complications after surgery in elderly patients, affecting between 20 and 40% of patients older than 60 after major surgery. This complication has huge consequences for the patients, families and society: increase of morbidity and mortality, prolonged length of stay, cognitive and functional decline leading to loss of autonomy, and important additional healthcare costs.

Among numerous risk factors identified, perioperative inflammatory stress is a key element in delirium genesis: surgical trauma releases danger signals in systemic circulation, activating immune cells and leading to neuroinflammation.

Melatonin is a neurohormone regulating circadian rhythm. But it also exhibits antioxidant and free radical scavenger properties, and regulates energy metabolism and immune function. It has already demonstrated a neuroprotective potential in various animal models. Its use against delirium is promising: it decreases delirium incidence in elderly patients hospitalized in medical ward, and several studies are now recruiting in ICU.

The hypothesis of the trial is that in a high-risk population, perioperative melatonin can reduce the incidence of POD.

The main objective is to evaluate the effect of perioperative melatonin administration on postoperative delirium incidence in the first 10 days after surgery, in elderly patients (over 70 years old) being hospitalized and scheduled for acute surgery of fractured lower limb (from femoral head to tibial plateau).

This is a prospective, national multicentric (24 centers), phase III, superiority, comparative randomized (1:1) double-blinded clinical trial with two parallel arms:

Experimental group: melatonin 4mg per os every night, starting the evening before surgery (or 2 hours before emergency surgery) and until day 5 after surgery.

Control group: placebo of this drug with the same schedule, during the same period of time.

The patients are aged 70 or older, hospitalized and scheduled for surgery of a severe fracture of a lower limb (from femoral head to tibial plateau).

DETAILED DESCRIPTION:
Postoperative delirium (POD) is one of the most frequent complications after surgery in elderly patients, affecting between 20 and 40% of patients older than 60 after major surgery. This complication has huge consequences for the patients, families and society: increase of morbidity and mortality, prolonged length of stay, cognitive and functional decline leading to loss of autonomy, and important additional healthcare costs.

Among numerous risk factors identified, perioperative inflammatory stress is a key element in delirium genesis: surgical trauma releases danger signals in systemic circulation, activating immune cells and leading to neuroinflammation. In the brain, especially in hippocampus, proinflammatory cytokines, immune cells recruitment and microglial activation alter synaptic plasticity and lead to acute cognitive dysfunction. Moreover, with aging, an increase in initial neuroinflammatory response and a decrease in subsequent resolution phase are observed.

Melatonin is a neurohormone regulating circadian rhythm. But it also exhibits antioxidant and free radical scavenger properties, and regulates energy metabolism and immune function. It has already demonstrated a neuroprotective potential in various animal models. Its use against delirium is promising: it decreases delirium incidence in elderly patients hospitalized in medical ward, and several studies are now recruiting in ICU. Concerning the perioperative period, only two studies with conflicting results are available. The first one (Sultan, 2010), that has shown that melatonin decreases POD incidence, has strong methodological limitations (no calculated sample size, only 53 patients in melatonin group, all patients, even in the control group received melatonin if they developed POD, etc). In the second one (deJonghe, 2014), melatonin had no effect on POD incidence, but showed a reduction in the proportion of patients with POD exceeding 2 days. These conflicting results emphasize the need for a third RCT, with optimized methodology.

The hypothesis of the trial is that in a high-risk population, perioperative melatonin can reduce the incidence of POD.

The main objective is to evaluate the effect of perioperative melatonin administration on postoperative delirium incidence in the first 10 days after surgery, in elderly patients (over 70 years old) being hospitalized and scheduled for acute surgery of fractured lower limb (from femoral head to tibial plateau).

This is a prospective, national multicentric (24 centers), phase III, superiority, comparative randomized (1:1) double-blinded clinical trial with two parallel arms:

Experimental group: melatonin 4mg per os every night, starting the evening before surgery (or 2 hours before emergency surgery) and until day 5 after surgery.

Control group: placebo of this drug with the same schedule, during the same period of time.

The patients are aged 70 or older, hospitalized and scheduled for surgery of a severe fracture of a lower limb (from femoral head to tibial plateau).

An ancillary study is also planned in this study with the hypothesise that :

* Patients presenting post-operative delirium may exhibit significant perturbations of phenotypic and transcriptomic features of circulating leukocytes, of plasma levels of cytokines, and of oxidative stress level.
* Administration of melatonin may prevent these perturbations.

Ancillary study concerns Beaujon, Bichat and la Pitié centers.

ELIGIBILITY:
Inclusion Criteria:

* Demographic criteria: patient 70 years old or older
* Diagnostic criteria: isolated fracture of a lower limb

  * Proximal femoral fractures: head, cervical, or trochanteric fractures
  * Periprosthetic hip fracture
  * Femoral shaft fracture
  * Distal femoral fractures: supracondylar or condylar
  * Periprosthetic knee fracture
  * Tibial plateau fracture
* Treatments/strategies/procedures: scheduled orthopedic surgery (osteosynthesis or arthroplasty)
* proxy or care giver knowing baseline cognitive status of the patient present or reachable by phone for an interview

Exclusion Criteria:

* Patient already taking Melatonin
* Contraindications and precaution for use of Melatonin administration:

  * Hypersensitivity to the active substance or to any of the excipients of Circadin©
  * Liver failure (presence of some of the following clinical and biological symptoms: icterus, asterixis, ascites, known esophageal varices, total bilirubin >20 micromol/L, FV <70%),
  * Cirrhosis (known histological liver fibrosis)
  * Renal failure with clearance <30 ml/min O Autoimmune disease O Hereditary galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption syndrome
  * Patients taking fluvoxamine, 5- or 8-methoxypsoralen, cimetidine, oestrogenotherapy, quinolones, carbamazepine, rifampicin
* Other concomitant trauma than lower limb fracture(s)
* Surgery scheduled in more than 5 days
* Patient under mechanical ventilation
* Patient refusing to participate
* Patient not talking / understanding French (delirium assessment impossible)
* Patient already participating to another interventional study
* No signed informed consent,
* No affiliation to a social security regime

Secondary Exclusion Criteria:

Secondary exclusion (before randomization): diagnosis of delirium at the CAM assessment at inclusion, or creatinin clearance <30 ml / min and /or biological signs of hepatocellular insufficiency (bilirubin> 20 umol/l and factor V <70%) if samples not available during the anesthesiologist consultation and so performed after inclusion.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 357 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium incidence | 10 days after surgery
  The Confusion Assessment Method (CAM) score, for patients hospitalized in surgery, or CAM-ICU score, for patients hospitalized in ICU will be applied daily during the first 10 days after surgery or end of hospital stay if shorter

SECONDARY OUTCOMES:
Number of days CAM positive | 10 days after surgery
  CAM will be applied daily during the first 10 days. the minimum 0 and maximum 4 values, and higher scores mean a worse outcome.
Incidence of postoperative sedative or antipsychotic drugs administration from | 10 days after surgery
  Daily review of the medical chart and prescriptions looking for any sedative or antipsychotic drug administration
Incidence of postoperative physical restrain prescription | 10 days after surgery
  Daily review of the medical chart and prescriptions looking for physical restraint prescription.
Incidence of postoperative falls | 10 days after surgery
  Daily review of the medical chart and prescriptions looking for falls, whichever the gravity
Mini Mental State Examination | 10 days (or end of hospital stay if shorter)
  Cognitive testing interview at bedside using the widely used French validated translation of the Mini Mental State Examination.
  the minimum 0 and maximum 30 values, and higher scores mean a better outcome.
Duration of hospital stay | 30 days after surgery
  Daily review of the medical file
30 days postoperative mortality | 30 days after surgery
  Phone call (or visit for those who had not left the hospital) to the patient or caregivers
30 days postoperative patient autonomy | 30 days after surgery
  Phone call (or visit for those who had not left the hospital) to the patient or caregivers and evaluation by the Katz Index of activities of daily living.
  The minimum and maximum values are respectively 0 and 6, and higher scores mean a better outcome.
30 days postoperative Quality of life | 30 days after surgery
  evaluated by EQ5D5L (standardized instrument for measuring generic health status : MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN/DISCOMFORT and ANXIETY/ DEPRESSION),) Questionnaire. the minimum 5 and maximum 125 values, and higher scores mean a better outcome.
30 days postoperative QALYs (quality-adjusted life year) | 30 days after surgery
  QALYs (quality-adjusted life year) are the utility weights for the 30 day period x30/365. the minimum and maximum values are respectively 0 and1, and higher scores mean a better outcome.
Total hospital costs at 30 days | 30 days after surgery
  calculated as the cumulative costs of all admissions (in- and outpatient, home care, rehabilitation) over a 30 day period
Incremental cost effectiveness | 30 days after surgery
  The incremental cost effectiveness ratio is the difference in total costs divided by the difference in the incidence rate of delirium between the two arms
cost utility ratios | 30 days after surgery
  the incremental cost utility ratio is the difference in total costs divided by the difference in QALYs (quality-adjusted life year)
Occurrence of side effects | 30 days after surgery
  During the follow-up, daily interview of the patient and review of the medical chart will be performed, looking for side effects of melatonin.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Sigaut, Principal Investigator — APHP
Locations (1):
- hôpital Beaujon, Clichy-sous-Bois, France

REFERENCES:
- [Derived] Sigaut S, Couffignal C, Esposito-Farese M, Degos V, Molliex S, Boddaert J, Raynaud-Simon A, Durand-Zaleski I, Marcault E, Jacota M, Dahmani S, Paugam-Burtz C, Weiss E. Melatonin for prevention of postoperative delirium after lower limb fracture surgery in elderly patients (DELIRLESS): study protocol for a multicentre randomised controlled trial. BMJ Open. 2021 Dec 24;11(12):e053908. doi: 10.1136/bmjopen-2021-053908. PMID 34952881